CLINICAL TRIAL: NCT03118674
Title: Newer Direct-Acting Anti-Viral Agents as Sole Therapy of Porphyria Cutanea Tarda in Subjects With Chronic Hepatitis C
Brief Title: Harvoni Treatment Porphyria Cutanea Tarda
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Gilead Sciences (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00043341; U54DK083909 (NIH)
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-05

CONDITIONS: Porphyria Cutanea Tarda; Hepatitis C
Keywords: Interventional, Open-label, PCT, Hepatitis C
MeSH Terms: conditions — Porphyria Cutanea Tarda; Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination; ledipasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Harvoni (Experimental): 1 tablet per day, oral, taken with or without food. 8 weeks for patients without cirrhosis, not previously treated with HCV GT1 and HCV rNA < 6 million IU/mL; 12 weeks for patients without cirrhosis; 24 weeks for patients with compensated cirrhosis
  Interventions: Drug: Harvoni

INTERVENTIONS:
Drug: Harvoni — One capsule of Harvoni/ ledipasvir, 90 mg + sofosbuvir, 400 mg administered daily for 8, 12, or 24 weeks
  Other Names: ledipasvir, 90 mg + sofosbuvir, 400 mg

SUMMARY:
In the medical literature there case reports that Harvoni improves symptoms in patients with PCT. However, this has never been systematically tested. Therefore, the purpose of this study is to assess whether Harvoni alone is an effective therapy of active PCT in patients with Chronic Hepatitis C.

DETAILED DESCRIPTION:
This is a clinical trial, which means its purpose is to study an intervention or treatment. In this study all patients with PCT will be given a standard dose of Harvoni and monitored for two years. Currently there are two standard therapies for PCT, phlebotomies (removing certain amounts of blood at specific intervals), or low dose hydroxychloroquine (an oral pill). These treatments are used for patients with PCT whether or not they also have HCV. For patients with HCV however, we do not know whether treating the HCV first will also resolve the PCT symptoms. There will be an initial visit to determine whether participants are eligible to be in the study. If a participant is found to be eligible, he/she will be asked come to the study site once every month over the course of one year, and then once every 3 months for an additional year. There will be approximately 17 visits over the course of the whole study. At these visits the study doctors will check in with the participant and some blood and urine samples will be taken. Participants will not be charged for any of the lab tests that are being done as a part of this study alone. All participants in this study will receive the Harvoni pills at no cost to them.

ELIGIBILITY:
Inclusion Criteria

1. Willing and able to give informed consent
2. ≥18 years of age
3. Symptoms and signs consistent with PCT and well documented biochemical diagnosis (urinary total porphyrin excretion > 500 mcg/g Creatinine with HPLC pattern typical of PCT-predominance of 8- and 7-carboxyl porphyrins)
4. Clinical diagnosis of PCT established by a study PI
5. Chronic hepatitis C: HCV RNA positive and quantifiable in serum detected within 90 days of enrollment, and documented HCV genotypes 1,4, 5, or 6 for which Harvoni is an approved therapy.
6. Women of child-bearing potential must be willing to avoid pregnancy and use an accepted and effective contraceptive method during treatment.

Exclusion Criteria

1. Women who are pregnant or who are breast-feeding
2. Patients who have already started treatment of PCT with phlebotomy or low dose hydroxychloroquine or chloroquine, or who have been in such treatment in the past 30 days
3. Patients who have already started another treatment regimen for CHC, or who have taken such treatment in the past 30 days
4. HIV infection with CD4 counts at baseline less than 350/µL or with evidence of any active AIDS-defining illnesses
5. Ongoing active alcohol abuse, defined as a history of drinking more than 25 drinks of alcohol per week during most weeks in the prior 4 months (History of prior, but not current alcohol abuse will NOT be grounds for exclusion because we seek to treat subjects with PCT and CHC of the type typically seen in clinical practice)
6. Any ongoing active IV drug use
7. Patients who are taking amiodarone or who have taken amiodarone within 60 days prior to enrollment
8. Patients who are taking, or within the prior 28 days have taken, rifampicin or St John's wort (Hypericum perforatum), both of which are P-gp inducers, which may significantly reduce the drug levels and therapeutic effects of Harvoni
9. Uncontrolled diabetes (Hgb A1c >9.5% within 60 days prior to enrollment)
10. Chronic hepatitis B
11. Autoimmune hepatic liver injury-autoimmune hepatitis, primary biliary cholangitis/sclerosing cholangitis or overlap syndrome
12. Alcoholic hepatitis
13. Other metabolic disorders of the liver, e.g. Alpha 1 antitrypsin deficiency with ZZ Pi type, Wilson's disease
14. Prior known or suspected drug-induced liver injury within 6 months of enrollment
15. Known or suspected hepatocellular carcinoma
16. On liver transplant list, or current MELD >12
17. History of liver transplant
18. Estimated GFR (Creatinine clearance) <30 mL/min (per Sofosbuvir being cleared by the kidney)
19. Serum ALT or AST >10x normal
20. Serum bilirubin >2 mg/dL (excluding patients with known or suspected Gilbert's syndrome)
21. Any other comorbid condition, which, in the opinion of the investigator, precludes participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L Bonkovsky, MD, Study Chair — Wake Forest University Health Sciences; Sean Rudnick, MD, Study Director — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonkovsky HL, Rudnick SP, Ma CD, Overbey JR, Wang K, Faust D, Hallberg C, Hedstrom K, Naik H, Moghe A, Anderson KE. Ledipasvir/Sofosbuvir Is Effective as Sole Treatment of Porphyria Cutanea Tarda with Chronic Hepatitis C. Dig Dis Sci. 2023 Jun;68(6):2738-2746. doi: 10.1007/s10620-023-07859-8. Epub 2023 Feb 22. PMID 36811718
- See also: Porphyrias Consortium Website — http://www.rarediseasesnetwork.org/cms/porphyrias/Studies

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Harvoni
Started | 23
Completed | 8
Not Completed | 15
Not completed — Lost to Follow-up | 2
Not completed — Screen Faliure | 8
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: Participants that started treatment
Arm/Group | Harvoni
Number analyzed (Participants) | 15
Age, Continuous [Median (Standard Deviation); unit: years] | 58.9 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Resolution of Active PCT by 7 Months After Start of Therapy
Description: Resolution of active PCT, defined as normalization of plasma porphyrins (less than 0.9 mcg/dL) by 7 months after start of therapy
Time Frame: 7 months
Population: 9 observations collected at 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Harvoni
Number analyzed (Participants) | 9
Participants | 9

2. Secondary Outcome: Time to Resolution of Active PCT
Description: Time to resolution of active PCT, defined as cessation of any new blisters or bullae and normalization of plasma porphyrins
Time Frame: through study completion, an average of 1 year
Population: Observations for 6 participants collected at through study completion, an average of 1 year
Measure: Mean (Full Range); unit: days
Arm/Group | Harvoni
Number analyzed (Participants) | 6
days | 240 [100 to 615]

3. Secondary Outcome: Number of Participants With Complete Biochemical Remission of PCT
Description: Defined as a decrease of the sum of urinary uro- and hepta-carboxyl porphyrins to less than 100 mcg/g creatinine and a normal urine porphyrin HPLC pattern defined as the total of highly carboxylated porphyrins (uro- and heptacarboxyl-porphyrins) being less than that of coproporphyrins, and the absence of a plasma fluorescence peak by fluorescence scanning
Time Frame: 12 Months
Population: 6 Observations collected at 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Harvoni
Number analyzed (Participants) | 6
Participants | 5

4. Secondary Outcome: Number of Participants With Cure of CHC
Description: Defined as no detectable HCV RNA at end of treatment and persisting for at least 12 weeks after end of treatment.
Time Frame: Up to 15 months
Population: 2 participants lost of follow up, 1 participant left the study after 4 weeks of dosing
Measure: Count of Participants; unit: Participants
Arm/Group | Harvoni
Number analyzed (Participants) | 12
Participants | 11

ADVERSE EVENTS:
Time Frame: Baseline through study completion, an average of 1 year
Arm/Group | Harvoni
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harvoni (N=15)
Hypertension (Vascular disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus pressure (General disorders) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (General disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in both hands (Musculoskeletal and connective tissue disorders) | 1 (1) — extreme pain in both hands due to PCT
Skin infection (Infections and infestations) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
We were not able to recruit as many subjects as we had originally planned and hoped to enroll [original target n = 49].

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT03118674/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT03118674/ICF_000.pdf